CLINICAL TRIAL: NCT00308581
Title: Phase IIIb Open-label Induction and Double-blind Comparison of 2 Maintenance Schedules Evaluating Clinical Benefit and Tolerability of Certolizumab Pegol in Crohn's Disease Patients With Prior Loss of Response or Intolerance to Infliximab
Brief Title: Certolizumab in Crohn's Disease Patients With Loss of Response or Intolerance to Infliximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87042; Eudract number: 2005-004104-37
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2011-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Certolizumab pegol
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active 1 (Experimental): Q4W regimen
  - every 4 weeks: alternatively placebo and 400mg Certolizumab Pegol
  Interventions: Biological: Certolizumab pegol; Other: Placebo
- Active 2 (Experimental): Q2W regimen
  - every 2 weeks: 400 mg Certolizumab Pegol
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — 400mg Certolizumab Pegol, Q4W, administered 4-weekly
  Other Names: CDP870; Cimzia
  Arms: Active 1
Biological: Certolizumab pegol — 400mg Certolizumab Pegol, Q2W, administered 2-weekly
  Other Names: CDP870; Cimzia
  Arms: Active 2
Other: Placebo — placebo administered 4-weekly in Active 1
  Arms: Active 1

SUMMARY:
To assess the clinical efficacy of subcutaneous (sc) certolizumab pegol administration over 26 weeks in patients suffering from Crohn's Disease (CD) and previously treated with infliximab

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Crohn's Disease
* Previous treatment failure to Infliximab (intolerance and/or no response)

Exclusion Criteria:

* Obstructive intestinal strictures
* Recent bowel resection
* Proctocolectomy or total colectomy
* Current total parenteral nutrition
* Short bowel syndrome
* All concomitant diseases or pathological conditions that could interfere with Crohn's disease assessment or to be harmful for the well being of the patient
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (107):
- United States (31):
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Lincoln, Nebraska
  - Great Neck, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Austria (3):
  - Innsbruck
  - Oberpullendorf
  - Vienna
- Belgium (8):
  - Bonheiden
  - Brussels
  - Genk
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Richmond, Ontario
  - Toronto, Ontario
  - Calgary
- Denmark (4):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Herlev
- France (10):
  - Amiens
  - Clichy
  - Grenoble
  - Lille
  - Montpellier, Cédex 5
  - Nice
  - Paris
  - Pessac
  - Rouen
  - Toulouse
- Germany (9):
  - Berlin
  - Hamburg
  - Hanover
  - Herne
  - Kiel
  - Leipzig
  - Minden
  - Munich
  - München
- Italy (7):
  - Bari
  - Bologna
  - Milan
  - Padua
  - Palermo
  - Roma
  - Torino
- Netherlands (7):
  - Amsterdam
  - Eindhoven
  - Enschede
  - Heerlen
  - Leiden
  - Terneuven
  - Zwolle
- Norway (2):
  - Oslo
  - Tromsø
- Spain (6):
  - Barcelona
  - Madrid
  - Oviedo
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Malmo
  - Örebro
  - Stockholm
- Switzerland (3):
  - Basel
  - Bern
  - Lausanne
- United Kingdom (7):
  - Bristol
  - Cambridge
  - Edinburgh
  - London
  - Nottingham
  - Oxford
  - Sheffield

REFERENCES:
- [Background] Taylor P, Manger B, Alvaro-Gracia J, Johnstone R, Gomez-Reino J, Eberhardt E, Wolfe F, Schwartzman S, Furfaro N, Kavanaugh A. Patient perceptions concerning pain management in the treatment of rheumatoid arthritis. J Int Med Res. 2010 Jul-Aug;38(4):1213-24. doi: 10.1177/147323001003800402. PMID 20925993
- [Result] Sandborn WJ, Abreu MT, D'Haens G, Colombel JF, Vermeire S, Mitchev K, Jamoul C, Fedorak RN, Spehlmann ME, Wolf DC, Lee S, Rutgeerts P. Certolizumab pegol in patients with moderate to severe Crohn's disease and secondary failure to infliximab. Clin Gastroenterol Hepatol. 2010 Aug;8(8):688-695.e2. doi: 10.1016/j.cgh.2010.04.021. Epub 2010 May 6. PMID 20451663
- [Result] Feagan BG, Sandborn WJ, Wolf DC, Coteur G, Purcaru O, Brabant Y, Rutgeerts PJ. Randomised clinical trial: improvement in health outcomes with certolizumab pegol in patients with active Crohn's disease with prior loss of response to infliximab. Aliment Pharmacol Ther. 2011 Mar;33(5):541-50. doi: 10.1111/j.1365-2036.2010.04568.x. Epub 2011 Jan 12. PMID 21223344
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 539 subjects that have been enrolled in the induction phase, 373 have been included in the randomized maintenance phase. The Baseline Characteristics module only includes the Intent-to-treat (ITTI) population of the induction phase.
Groups:
- Q4W Regimen: every 2 weeks: alternatively placebo and 400 mg Certolizumab Pegol
- Q2W Regimen: every 2 weeks: 400 mg Certolizumab Pegol
- Overall: Overall Induction
Period: Induction Phase
Arm/Group | Q4W Regimen | Q2W Regimen | Overall
Started | 0 (Not applicable in this period) | 0 (Not applicable in this period) | 539
Completed | 0 (Not applicable in this period) | 0 (Not applicable in this period) | 373
Not Completed | 0 | 0 | 166
Not completed — Adverse Event | 0 | 0 | 37
Not completed — Lack of Efficacy | 0 | 0 | 121
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Unknown reason | 0 | 0 | 3
Period: Randomized Maintenance Phase
Arm/Group | Q4W Regimen | Q2W Regimen | Overall
Started | 187 | 186 | 0
Completed | 82 | 83 | 0
Not Completed | 105 | 103 | 0
Not completed — Adverse Event | 10 | 17 | 0
Not completed — Lack of Efficacy | 9 | 21 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Switched to Q2W open-label treatment | 82 | 59 | 0
Not completed — Unknown reason | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 526
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.67 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345
  Male | 194
Region of Enrollment [Number; unit: participants]
  United States | 141
  Spain | 11
  Austria | 16
  United Kingdom | 29
  Italy | 53
  Switzerland | 8
  France | 45
  Canada | 43
  Belgium | 88
  Denmark | 11
  Germany | 64
  Netherlands | 17
  Norway | 9
  Sweden | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Status With Response Defined as at Least 100 Point Decrease in Crohn's Disease Activity Score (CDAI Score) From Baseline in the Induction Phase
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score) from baseline, otherwise there is a non-response.
  The CDAI score is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline to Week 6
Population: Intent-to-treat Induction Phase (ITTI) population: subjects who received at least one dose of study drug in the induction phase
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 539
participants
  Response | 334
  Non-Response | 205

2. Secondary Outcome: Response Status With Response Defined as at Least 100 Point Decrease in CDAI Score From Baseline in the Randomized Maintenance Phase
Description: Response is defined as at least 100 point decrease in CDAI score from baseline. The CDAI score is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline to Week 26
Population: Intent-to-treat Randomized Maintenance Phase (ITTR) population: subjects who were randomized and received at least one dose of study drug in the randomized maintenance phase
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 187 | 186
participants
  Response | 70 | 66
  Non-Response | 117 | 120
Statistical Analysis 1: Comparison: Q4W Regimen vs Q2W Regimen; With a sample size of 165 patients per treatment arm, assuming a percentage of responders of 45% with the Q4W regimen, the study had 80% power to show a statistically significant difference in percentage of responders at Week 26 between the two treatment groups, when there is a true difference of 16% in percentage of responders in favor of the Q2W regimen, and using a 2-sided chi-square at the 5% significance level; Test type: Superiority or Other; p = 0.696, Regression, Logistic — Logistic regression model including terms for treatment arm and geographical region (North America versus Europe); Odds Ratio (OR) = 1.1, 95% CI [0.7 to 1.7] — Direction of comparison is Q4W regimen (active 1) versus Q2W regimen (active 2)

3. Secondary Outcome: Response Status With Response Defined as at Least 70 Points Reduction in CDAI Score in the Induction Phase
Description: Response is defined as at least 70 points reduction in CDAI score. The CDAI score is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline to Week 6
Population: ITTI population: all subjects who received at least one dose of study drug in the induction phase
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 539
participants
  Response | 373
  Non-response | 166

4. Secondary Outcome: Response Status With Response Defined as at Least 70 Points Reduction in CDAI Score in the Randomized Maintenance Phase
Description: as for outcome 3
Time Frame: Baseline to Week 26
Population: ITTR population: subjects who were randomized and received at least one dose of study drug in the randomized maintenance phase
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 187 | 186
participants
  Response | 75 | 75
  Non-response | 112 | 111

5. Secondary Outcome: Remission Status With Remission Defined as CDAI Score ≤ 150 in the Induction Phase
Description: Remission is defined as CDAI score ≤ 150. The CDAI score is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 6
Population: ITTI population: subjects who received at least one dose of study drug in the induction phase
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 539
participants
  Remission | 212
  No remission | 327

6. Secondary Outcome: Remission Status With Remission Defined as CDAI Score ≤ 150 in the Randomized Maintenance Phase
Description: Remission is defined as CDAI score ≤ 150. The CDAI score is used to quantify the symptoms with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 26
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 187 | 186
participants
  Remission | 51 | 52
  No remission | 136 | 134

7. Secondary Outcome: CDAI Score at Week 2 of the Induction Phase
Description: The CDAI score is used to quantify the symptoms of subjects with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 2
Population: ITTI population: all subjects who received at least one dose of study drug in the induction phase (available measurements)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 535
points on a scale | 241.53 (97.03)

8. Secondary Outcome: CDAI Score at Week 4 of the Induction Phase
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 522
points on a scale | 220.87 (101.05)

9. Secondary Outcome: CDAI Score at Week 6 of the Induction Phase
Description: as for outcome 7
Time Frame: Week 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 499
points on a scale | 187.81 (103.34)

10. Secondary Outcome: CDAI Score at Week 8 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 8
Population: ITTR population: subjects who were randomized and received at least one dose of study drug in the randomized maintenance phase (available measurements)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 184 | 181
points on a scale | 175.62 (94.08) | 169.18 (86.63)

11. Secondary Outcome: CDAI Score at Week 10 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 178 | 167
points on a scale | 164.65 (98.16) | 162.86 (88.66)

12. Secondary Outcome: CDAI Score at Week 12 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 161 | 153
points on a scale | 173.83 (103.89) | 163.78 (96.19)

13. Secondary Outcome: CDAI Score at Week 14 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 143 | 142
points on a scale | 162.34 (99.74) | 158.68 (90.76)

14. Secondary Outcome: CDAI Score at Week 16 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 129 | 131
points on a scale | 163.73 (103.65) | 156.05 (90.49)

15. Secondary Outcome: CDAI Score at Week 18 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 114 | 113
points on a scale | 153.38 (95.65) | 156.64 (90.99)

16. Secondary Outcome: CDAI Score at Week 20 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 20
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 104 | 98
points on a scale | 162.79 (112.53) | 138.60 (80.78)

17. Secondary Outcome: CDAI Score at Week 22 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 22
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 88 | 91
points on a scale | 128.13 (85.34) | 141.89 (90.43)

18. Secondary Outcome: CDAI Score at Week 24 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 82 | 85
points on a scale | 135.49 (99.92) | 139.50 (75.98)

19. Secondary Outcome: CDAI Score at Week 26 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Week 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 81 | 83
points on a scale | 122.37 (87.49) | 131.41 (79.52)

20. Secondary Outcome: Change From Baseline in CDAI Score at Week 2 of the Induction Phase
Description: as for outcome 7
Time Frame: Baseline to Week 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 534
points on a scale | -66.57 (85.73)

21. Secondary Outcome: Change From Baseline in CDAI Score at Week 4 of the Induction Phase
Description: as for outcome 7
Time Frame: Baseline to Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 521
points on a scale | -87.63 (93.89)

22. Secondary Outcome: Change From Baseline in CDAI Score at Week 6 of the Induction Phase
Description: as for outcome 7
Time Frame: Baseline to Week 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Overall
Number analyzed (Participants) | 498
points on a scale | -120.33 (90.81)

23. Secondary Outcome: Change From Baseline in CDAI Score at Week 8 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 184 | 181
points on a scale | -133.35 (85.90) | -137.70 (75.89)

24. Secondary Outcome: Change From Baseline in CDAI Score at Week 10 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 178 | 167
points on a scale | -145.16 (90.76) | -145.26 (76.97)

25. Secondary Outcome: Change From Baseline in CDAI Score at Week 12 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 161 | 153
points on a scale | -134.51 (91.52) | -145.17 (78.88)

26. Secondary Outcome: Change From Baseline in CDAI Score at Week 14 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 143 | 142
points on a scale | -145.54 (86.85) | -144.08 (86.34)

27. Secondary Outcome: Change From Baseline in CDAI Score at Week 16 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 129 | 131
points on a scale | -141.90 (98.56) | -144.89 (83.81)

28. Secondary Outcome: Change From Baseline in CDAI Score at Week 18 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 18
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 114 | 113
points on a scale | -150.38 (88.68) | -144.66 (85.43)

29. Secondary Outcome: Change From Baseline in CDAI Score at Week 20 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 20
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 104 | 98
points on a scale | -139.98 (104.52) | -162.85 (80.93)

30. Secondary Outcome: Change From Baseline in CDAI Score at Week 22 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 22
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 88 | 91
points on a scale | -171.52 (82.56) | -159.13 (88.94)

31. Secondary Outcome: Change From Baseline in CDAI Score at Week 24 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 82 | 85
points on a scale | -165.06 (90.54) | -160.44 (76.11)

32. Secondary Outcome: Change From Baseline in CDAI Score at Week 26 in the Randomized Maintenance Phase
Description: as for outcome 7
Time Frame: Baseline to Week 26
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 81 | 83
points on a scale | -176.85 (80.44) | -168.59 (77.03)

33. Other Pre Specified Outcome: Time to Loss of Response (CDAI Score > 150 and Minimum Increase in CDAI of 70) After Week 6
Description: Median time to loss of response in the maintenance period (from Kaplan-Meier analysis); range is time of first event to time of last event. Loss of response is defined as both a CDAI score > 150 points and a minimum increase in CDAI of 70 points versus Week 6 at two consecutive visits.
Time Frame: Week 6 to Week 26
Population: as for outcome 10
Measure: Median (Full Range); unit: days
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 168 | 161
days | 128 [10 to 133] | 125 [14 to 141]

34. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 10 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 10
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 2 | 2

35. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 12 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 12
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 3 | 4

36. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 14 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 14
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 3 | 3

37. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 16 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 16
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 5 | 8

38. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 18 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 18
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 7 | 7

39. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 20 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 20
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 8 | 6

40. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 22 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 22
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 8 | 7

41. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 24 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 24
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 9 | 5

42. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Remission at Week 26 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Remission is defined as CDAI score ≤ 150.
Time Frame: Week 26
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 8 | 5

43. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 10 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 10
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 2 | 2

44. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 12 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 12
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 4 | 4

45. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 14 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 14
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 5 | 5

46. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 16 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 16
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 8 | 10

47. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 18 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 18
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 9 | 8

48. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 20 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 20
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 9 | 7

49. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 22 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 22
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 9 | 8

50. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 24 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 24
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 11 | 5

51. Secondary Outcome: Number of Patients Able to Taper and Discontinue Steroids While Maintaining Response at Week 26 in the Randomized Maintenance Phase in the Subset of Patients Taking Steroids at Baseline.
Description: Response is defined as at least 100 point decrease in Crohn's Disease Activity Score (CDAI score).
Time Frame: Week 26
Population: ITTR population taking steroids at baseline
Measure: Number; unit: participants
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 76 | 78
participants | 10 | 6

52. Secondary Outcome: C - Reactive Protein (CRP) Level at Baseline (Week 0) of the Induction Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 0
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Overall
Number analyzed (Participants) | 529
mg/L | 9.5 [2.5 to 27.8]

53. Secondary Outcome: CRP Level at Week 2 of the Induction Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 2
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Overall
Number analyzed (Participants) | 528
mg/L | 4.2 [1.3 to 14.8]

54. Secondary Outcome: CRP Level at Week 4 of the Induction Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 4
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Overall
Number analyzed (Participants) | 514
mg/L | 3.8 [1.2 to 16.0]

55. Secondary Outcome: CRP Level at Week 6 of the Induction Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 6
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Overall
Number analyzed (Participants) | 493
mg/L | 4.2 [1.4 to 16.4]

56. Secondary Outcome: CRP Level at Week 8 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 8
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 182 | 181
mg/L | 5.6 [1.4 to 20.4] | 4.6 [1.2 to 15.8]

57. Secondary Outcome: CRP Level at Week 10 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 10 (optional measurement)
Population: ITTR population: subjects who were randomized and received at least one dose of study drug in the randomized maintenance phase (available measurements, measurements are optional)
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 0 | 4
mg/L |  | 5.3 [4.3 to 11.1]

58. Secondary Outcome: CRP Level at Week 12 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 158 | 149
mg/L | 5.4 [1.8 to 18.9] | 3.7 [1.3 to 14.1]

59. Secondary Outcome: CRP Level at Week 14 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 14 (optional measurement)
Population: as for outcome 57
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 1 | 1
mg/L | 0.6 [0.6 to 0.6] | 3.0 [3.0 to 3.0]

60. Secondary Outcome: CRP Level at Week 16 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 16
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 125 | 130
mg/L | 5.5 [1.8 to 19.4] | 4.4 [1.3 to 12.1]

61. Secondary Outcome: CRP Level at Week 18 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 18 (optional measurement)
Population: as for outcome 57
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 3 | 3
mg/L | 18.4 [3.4 to 110.2] | 5.9 [0.7 to 10.1]

62. Secondary Outcome: CRP Level at Week 20 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 20
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 100 | 97
mg/L | 6.8 [1.9 to 26.0] | 4.4 [1.6 to 13.7]

63. Secondary Outcome: CRP Level at Week 22 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 22 (optional measurement)
Population: as for outcome 57
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 0 | 2
mg/L |  | 13.0 [1.6 to 24.4]

64. Secondary Outcome: CRP Level at Week 24 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 24
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 82 | 83
mg/L | 5.2 [1.6 to 24.4] | 4.6 [1.7 to 13.2]

65. Secondary Outcome: CRP Level at Week 26 in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L.
Time Frame: Week 26
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 79 | 82
mg/L | 5.4 [1.6 to 17.0] | 5.1 [1.5 to 14.8]

66. Secondary Outcome: CRP Level at Endpoint (Last Visit) in the Randomized Maintenance Phase
Description: High CRP levels are defined as greater or equal 5 mg/L, normal or low levels are below 5 mg/L. Endpoint is the visit when the last observation was taken, either at week 26 or at a visit before in case of early dropout.
Time Frame: Last visit on or before Week 26
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Q4W Regimen | Q2W Regimen
Number analyzed (Participants) | 183 | 184
mg/L | 6.9 [1.9 to 22.4] | 4.8 [1.5 to 18.7]

ADVERSE EVENTS:
Time Frame: Adverse events are reported here for the induction phase + safety follow-up period following induction, and for the randomized maintenance phase + safety follow-up period following maintenance.
Groups:
- Q4W Regimen: Subjects who were randomized to and received Q4W regimen (every 2 weeks: alternatively placebo and 400 mg Certolizumab Pegol); randomized maintenance phase + safety follow-up period following randomized maintenance phase.
- Q2W Regimen: Subjects who were randomized to and received Q2W regimen (every 2 weeks: 400 mg Certolizumab Pegol); randomized maintenance phase + safety follow-up period following randomized maintenance phase.
- Induction Phase: Overall population in the Induction phase + safety follow-up period following induction phase.
Arm/Group | Q4W Regimen | Q2W Regimen | Induction Phase
Serious Adverse Events (participants affected / at risk) | 25/187 | 25/186 | 40/539
Other Adverse Events (participants affected / at risk) | 97/187 | 106/186 | 277/539
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q4W Regimen (N=187) | Q2W Regimen (N=186) | Induction Phase (N=539)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (4)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (5)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 10 (11) | 5 (5) | 23 (26)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Douglas' abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Obstruction (General disorders) | 0 (0) | 0 (0) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q4W Regimen (N=187) | Q2W Regimen (N=186) | Induction Phase (N=539)
Abdominal Pain (Gastrointestinal disorders) | 16 (18) | 18 (20) | 40 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (19) | 20 (22) | 51 (62)
Crohn's disease (Gastrointestinal disorders) | 8 (9) | 15 (15) | 21 (23)
Fatigue (General disorders) | 14 (15) | 10 (14) | 37 (40)
Headache (Nervous system disorders) | 31 (53) | 20 (21) | 86 (95)
Herpes simplex (Infections and infestations) | 11 (16) | 6 (9) | 8 (8)
Nasopharyngitis (Infections and infestations) | 23 (28) | 32 (35) | 41 (43)
Nausea (Gastrointestinal disorders) | 21 (27) | 20 (22) | 58 (65)
Pharyngolaryngeal pain (Reproductive system and breast disorders) | 12 (13) | 8 (10) | 20 (22)
Pyrexia (General disorders) | 20 (21) | 22 (25) | 46 (53)
Urinary tract infection (Infections and infestations) | 10 (12) | 7 (9) | 14 (14)
Vomiting (Gastrointestinal disorders) | 17 (17) | 12 (13) | 44 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.